CLINICAL TRIAL: NCT05116280
Title: Registration of the Major Adverse Cardiovascular Events and Pulmonary Embolism in Primary Total Joint Arthroplasty
Brief Title: MACE and PE in Elective Primary TKA & THA
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: MACE & PE in TJA
Record Dates: First submitted 2021-10-05; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Cardiovascular Complication; Pulmonary Embolism; Stroke; Transient Ischemic Attack; Death
Keywords: total joint arthroplasty; total hip arthroplasty; total knee arthroplasty; major adverse cardiovascular events; pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism; Stroke; Ischemic Attack, Transient; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TJA: patients with primary osteoarthritis of the knee and hip who underwent elective primary total hip and total knee arthroplasty.
  MACE and pulmonary embolism were recorded

SUMMARY:
This study ought to identify the occurence of the major adverse cardiovascular events (MACE) and the pumonary emoblism (PE) in patients undergoing elective primary THA & TKA

DETAILED DESCRIPTION:
The study included 220 consecutive patients undergoing elective primary THA & TKA from January 2018 to December 2018. The occcurence of major adverse cardiovascular events (MACE) and the pumonary emoblism (PE) were recorder. Under the term MACE the following were included; non fatal cardiac arrest acute myocardial infraction congestive cardiac failure cardiac arrhythmia agnina stroke cardiovascular death cerebrovascular death

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients age 18 years or older, with a diagnosis of primary osteoarthritis of the hip or knee, who underwent elective, primary, unilateral TKA or THA.

Exclusion Criteria:

* previous TKA or THA within 3 months
* Revision surgery
* Surgical procedures related to a previous complication
* ASA PS IV
* recent history (6 months) of unstable acute coronary syndrome or decompensated heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients age 18 years or older, with a diagnosis of primary osteoarthritis of the hip or knee, who underwent elective, primary, unilateral TKA or THA. Operations were performed by the 4 chief arthroplasty surgeons of the department.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 1month postoperatively
  MACE (non-fatal-cardiac arrest, acute myocardial infraction, congestive cardiac failure, cardiac arrhythmia, angina, stroke, cardiovascular death, cerebrovascular, death)
Pulmonary Embolism | 1month postoperatively
  PE

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Larissa, Greece